CLINICAL TRIAL: NCT06299839
Title: A Phase 1 Open-label Study to Assess the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of PAS-004, a MEK (1/2) Inhibitor, in Patients With MAPK Pathway-driven Advanced Solid Tumors With a Documented RAS, NF1, or RAF Mutation or Patients Who Have Failed BRAF/MEK Inhibition
Brief Title: PAS-004 in Patients With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Pasithea Therapeutics Corp. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PAS-004-102; 2024-510900-34 (EudraCT Number)
Record Dates: First submitted 2024-02-12; First posted 2024-03-08 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: RAS Mutation; NF1 Mutation; RAF Mutation; Advanced Solid Tumors
Keywords: Cancer; malignant neoplasms; Advanced Solid Tumors; MAP Kinase Signaling Pathway
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: 3+3 dose expansion
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- PAS-004 Capsules (Experimental): Sequential dose escalation: 2 mg, 4 mg, 8 mg, 15 mg, 22 mg, 30 mg, 37 mg, and 45 mg
  Interventions: Drug: PAS-004 Capsules
- PAS-004 Tablets (Experimental): A single cohort at the 4mg dose using tablet formulation of PAS-004
  Interventions: Drug: PAS-004 Tablets

INTERVENTIONS:
Drug: PAS-004 Capsules — A mitogen-activated protein kinase/extracellular signal-regulated kinase kinase (MAPK/ERK kinase, or MEK) 1/2 inhibitor presented in 1 mg, 4mg, and 10 mg strength capsules, intended for oral administration once daily.
  Arms: PAS-004 Capsules
Drug: PAS-004 Tablets — A mitogen-activated protein kinase/extracellular signal-regulated kinase kinase (MAPK/ERK kinase, or MEK) 1/2 inhibitor presented in 4mg strength tablets, intended for oral administration once daily.
  Arms: PAS-004 Tablets

SUMMARY:
The main purpose of this clinical trial is to test PAS-004 in people with advanced solid tumors with rat sarcoma virus (RAS), neurofibromatosis type I (NF1), or rapidly accelerated fibrosarcoma (RAF) mutations. The main questions it aims to answer are:

* How well participants are able tolerate different doses of PAS-004, and
* What side effects PAS-004 might have.

Study participants will have regular visits to the study doctor and be asked to have tests and exams done to check on their health and safety. Everyone participating in the study will take PAS-004 by mouth as a single dose, followed by one week observation, then once a day during the study, in 28-day cycles. Participants will continue on daily PAS-004 for up to 2 years, or until:

* They decide to withdraw from the study, or
* They experience unacceptable side effects, or
* Their disease progresses, or another illness interferes with taking the study drug, or
* The sponsors stops the study.

ELIGIBILITY:
Inclusion Criteria:

1. Capable of giving signed informed consent which includes compliance with the requirements, prohibitions and restrictions listed in the informed consent form (ICF).
2. Patient has been informed both verbally and in writing about the objectives of the clinical study, the methods, the anticipated benefits, the potential risks, and the discomfort to which they may be exposed and has given written consent to participation in the study prior to study start and any study-related procedure.
3. Patient must be at least 18 years of age at the time of signing the ICF.
4. Patient must be able to swallow oral medication.
5. Patient with histologically or cytologically diagnosed mitogen-activated protein kinase (MAPK) pathway driven advanced solid tumors with all of the following characteristics:

   1. Tumor cannot be surgically resected
   2. Patient has failed or is ineligible for standard of care therapy
   3. Patient has no available treatment options with known clinical benefit
   4. Documented evidence of rat sarcoma virus (RAS), neurofibromatosis type I (NF1), and/or rapidly accelerated fibrosarcoma (RAF) mutations. Patients with RAF mutations must have previously failed v-Raf murine sarcoma viral oncogene homolog B (BRAF) / MEK inhibition.
6. Prior to enrollment, patients without an existing prior genetic test result or adequate tumor tissue sample must agree to provide tumor tissue via biopsy (paraffin section or fresh tissue specimens) that will be sent for analysis to confirm eligibility.
7. Patient must have an Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1 (Appendix B).
8. Patient must have an estimated life expectancy of at least 12 weeks in the opinion of the Investigator at the time of informed consent.
9. Patient must have adequate organ function at screening as indicated by the following laboratory value ranges:

   1. Serum total bilirubin ≤ 1.5 × upper limit normal (ULN) (Serum total bilirubin can be ≤ 3.0 × ULN if patients have hemolysis or congenital hemolytic diseases)
   2. Aspartate aminotransferase (AST) ≤ 2.5 × ULN or 5 × ULN for patient with liver metastases
   3. Alanine aminotransferase (ALT) ≤ 2.5 × ULN or 5 × ULN for patient with liver metastases
   4. Albumin ≥2 mg/dL
   5. Creatinine clearance ≥ 45 mL/min (as calculated per Cockcroft-Gault)
   6. Absolute neutrophil count (ANC) ≥ 1.5×109/L
   7. Platelets ≥ 100×109/L
   8. Hemoglobin ≥ 90 g/L (Note: Criteria must be met without a transfusion within 2 weeks of obtaining the sample)
10. Patient must agree to maintain abstinence (no heterosexual intercourse) or use a highly effective form of contraception during study treatment and for at least 90 days after the last dose of IP. Male patients must agree not to donate sperm while receiving IP and for at least 90 days after the last dose of IP.

Exclusion Criteria:

1. Participation in another therapeutic clinical trial within 3 weeks of enrollment.
2. Having received chemotherapy, radiotherapy, major surgery, targeted therapy, immunotherapy, or other antitumor treatment within 21 days of enrollment or five half-lives of the administered therapy, whichever occurs first.
3. Known or active central nervous system metastases.

   1. Patients with untreated brain metastases ≤ 30 mm that are asymptomatic, do not have significant edema, and do not require steroids or anti-seizure medications are eligible after discussion with the Medical Monitor.
   2. Patients with previously treated brain metastases may participate provided they are stable after treatment and without evidence of progression by imaging for at least 4 weeks prior to the first dose of IP administration and are not using corticosteroids for at least 7 days prior to IP administration.
   3. Patients with confirmed leptomeningeal disease are to be excluded.
4. Unresolved toxicity from prior antitumor therapy defined as AEs > Grade 2 according to Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0, except for alopecia; neurotoxicity AEs of patients who have received prior chemotherapy needs to be restored to Grade 2 or below. Patients with ≥ Grade 3 bleeding within 4 weeks of first study treatment dose should be excluded.
5. Taken a medication that is a strong cytochrome P450 (CYP3A) inhibitor or inducer within 14 days of initiation of study therapy dosing.
6. Taken a known corrected QT (QTc) interval prolongating medication within 7 days of initiation or longer if the half-life of the QTc prolonging medication is such that the drug is not cleared from the body within 7 days (5 half-lives) of initiation of study therapy dosing.
7. Active dysphagia, digestive system disease, malabsorption syndrome, or other conditions affecting PAS-004 absorption.
8. Previous or current retinal vein stenosis, retinal detachment, central retinal vein occlusion, or currently active glaucoma.
9. Active interstitial pneumonia, including clinically significant radiation pneumonitis.
10. Impaired cardiac function or cardiac disease as indicated by:

    1. Average QTc interval > 470 ms as calculated according to the QTc formula of the instrument at the research center where electrocardiogram (ECG) measurements are performed.
    2. Grade ≥ 3 congestive heart failure per New York Heart Association (NYHA) guidelines.
    3. Clinically significant arrhythmias, including but not limited to, complete left bundle branch conduction abnormalities and 2nd degree atrioventricular block.
11. Pregnant or lactating female patients.
12. Known allergy or hypersensitivity to the investigational product (IP), including excipients, or history of severe adverse reaction to any drug, or sensitivity to components of the IP.
13. Clinically active bacterial, fungal, or viral infections, hepatitis B (hepatitis B virus surface antigen positive and hepatitis B virus DNA over 1000 IU/ml) or hepatitis C (hepatitis C virus RNA positive), human immunodeficiency virus infection (HIV positive).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2024-02-29 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Evaluation of dose limiting toxicities (DLTs) | Day 1 through Day 35 (Cycle 1)
  Pre-defined DLTs will be assessed for dose escalation and expansion determinations.
Evaluation of adverse events (AEs) | Screening through Day 1 through Day 35 (Cycle 1), and 30 days after discontinuation of study drug
  The number and severity of AEs will be evaluated for dosing cohorts to inform dose escalation and expansion decisions, and support selection of a preliminary recommended phase 2 dose (RP2D).
Evaluation of AEs leading to discontinuation of investigational product (IP), PAS-004. | Screening through Day 1 through Day 35 (Cycle 1), and 30 days after discontinuation of study drug
  The number and severity of AEs leading to discontinuation of study drug will be evaluated for dosing cohorts to inform dose escalation and expansion decisions, and support selection of a preliminary recommended phase 2 dose (RP2D).
Evaluation of hematology laboratory parameters | Screening through Day 1 through Day 35 (Cycle 1), and 30 days after discontinuation of study drug
  Lab parameters will be evaluated for to assess the safety profile of the study drug, and support selection of a preliminary recommended phase 2 dose (RP2D).
Evaluation of clinical chemistry laboratory parameters | Screening through Day 1 through Day 35 (Cycle 1), and 30 days after discontinuation of study drug
  Lab parameters will be evaluated for to assess the safety profile of the study drug, and support selection of a preliminary recommended phase 2 dose (RP2D).

SECONDARY OUTCOMES:
Apparent terminal elimination half-life (t1/2) in Plasma | Cycle 1: Day 1 and Day 22 (predose, and 30 min, 1 hr, 2 hr, 3 hr, 5 hr, 8 hr and 24 hr post-dose), Day 4, 8, 15, 29 and 35 (predose)
Peak Plasma Concentration (Cmax) | Cycle 1: Day 1 and Day 22 (predose, and 30 min, 1 hr, 2 hr, 3 hr, 5 hr, 8 hr and 24 hr post-dose), Day 4, 8, 15, 29 and 35 (predose)
Plasma predose or trough concentration (Ctau/Ctrough) | Cycle 1: Day 22 (predose, and 30 min, 1 hr, 2 hr, 3 hr, 5 hr, 8 hr and 24 hr post-dose), Day 8, 15, 29 and 35 (predose)
Time of maximum plasma concentration (Tmax) | Cycle 1: Day 1 and Day 22 (predose, and 30 min, 1 hr, 2 hr, 3 hr, 5 hr, 8 hr and 24 hr post-dose), Day 4, 8, 15, 29 and 35 (predose)
Area under the concentration versus time curve from time zero to the last sampling time with quantifiable analyte (AUC0-t) | Cycle 1: Day 1 (predose, and 30 min, 1 hr, 2 hr, 3 hr, 5 hr, 8 hr and 24 hr post-dose), Day 4
Area under the concentration versus time curve from time zero extrapolated to infinity if possible (AUC0-∞) | Cycle 1: Day 1 (predose, and 30 min, 1 hr, 2 hr, 3 hr, 5 hr, 8 hr and 24 hr post-dose), Day 4
Area under the concentration versus time curve for the dosing interval, assuming steady state has been reached and duplicating the predose concentration for the 24 hour postdose concentration (AUC0-tau) | Cycle 1: Day 22 (predose, and 30 min, 1 hr, 2 hr, 3 hr, 5 hr, 8 hr and 24 hr post-dose), Day 8, 15, 29 and 35 (predose)
Apparent total plasma clearance if possible (CL/F) | Cycle 1: Day 1 (predose, and 30 min, 1 hr, 2 hr, 3 hr, 5 hr, 8 hr and 24 hr post-dose), Day 4, and 8 (predose)
Evaluation of the percentage of extracellular signal-regulated kinase phosphorylation (pERK) inhibition from baseline | Day 1 through Day 35 (Cycle 1)
Evaluation of the objective response rate (ORR) | Screening, Day 35 (Cycle 1), and every 9 weeks thereafter
  The proportion of participants achieving a partial response (PR) or complete response (CR) per response evaluation criteria in solid tumors (RECIST) 1.1 criteria.
Evaluation of progression-free survival (PFS) | Cycle 1 Day 1 to date of death, up to 25 months from last participant enrolled
  The time from first dose of IP to the date of documented disease progression or date of death due to any cause (whichever occurs first).
Evaluation of overall survival (OS) | Cycle 1 Day 1 to date of death, up to 13 months from last participant enrolled
  The time from first dose of IP to the date of death due to any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Tiago R Marques, MD, Study Director — Pasithea Therapeutics Corp.
Locations (7):
- United States (4):
  - NEXT Oncology, Austin, Texas
  - NEXT Oncology, Irving, Texas
  - NEXT Oncology, San Antonio, Texas
  - NEXT Oncology, Fairfax, Virginia
- MBAL Sveta Sofia, Sofia, Bulgaria
- Romania (2):
  - Institute of Oncology Bucharest Prof. Dr. Alexandru Trestioreanu, Bucharest
  - Institute of Oncology Prof. Dr. Ion Chiricuta, Cluj-Napoca

IPD SHARING:
Plan to Share IPD: No